CLINICAL TRIAL: NCT01344577
Title: Buccal Plate Augmentation Associated With Different Hydroxyapatite-based Biomaterials. A Multicenter Randomized Controlled Clinical Trial
Brief Title: Buccal Plate Augmentation With Different Hydroxyapatite Based Material
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, chiara navarra, doctor, University of Trieste
Other Study IDs: BPA-2011-units
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Edentulous
Keywords: Buccal Plate Augmentation technique; socket preservation; porcine biomaterial
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group1#: bone graft material used: Apatos Cortical® (porcine cortical bone 600-1000 µm)
- Group2#: bone graft material used: MP3® (porcine cortic-cancellous collagenated bone mix 600-1000 µm)
- Group3#: control group

SUMMARY:
The purposes of this study are : (first) to evaluate comparatively the effectiveness of 2 HA-based biomaterials when used for socket preservation with Buccal Plate Augmentation technique; (second) to evaluate clinical outcomes of socket preservation procedures performed using the Buccal Plate Augmentation technique.

DETAILED DESCRIPTION:
Tooth loss results physiologically in a significant remodeling of the alveolar ridge. The bone resorption process begins immediately after extraction, leading to an average 40-60% decrease in the horizontal and vertical dimensions of the alveolar ridge, during the first 2 years (Amler 1969, Johnson 1969)1,2. The majority of post-extraction bone loss is more evident on the buccal aspect of the ridge (Pietrokovski & Massler 1967)3 and occurs mainly within the first 3 months (Johnson 1969; Schropp et al. 2003)2,4. It is now known that crestal remodeling is strictly related to bundle bone resorption5 and that is more evident on the buccal plate where, especially in thin periodontal biotypes, can result in significant facial hard and soft tissue recessions. Bundle bone vascularization comes from periodontal ligament and it is interrupted by tooth extraction: for this reason bundle bone resorption and, consequent socket remodeling are impossible to prevent. Furthermore, modeling and remodeling of extraction sockets have a great variability in timing: a recent study (Trombelli et al. 2008) reports that bone organization and architecture is not completed 24 weeks after tooth extraction6.

In order to preserve ridge volumetry after extraction, many clinical techniques and various biomaterials have been suggested for grafting of post-extraction wounds7-12. Grafting of sockets provides stable clinical results but some studies demonstrate that, unless using a membrane, at histological examination most of the graft particles are encapsulated by fibrous tissue, especially in the coronal area 9,11. Recently, a study on an animal model (Araújo et al. 2009) reported that the presence of bone graft material in fresh extraction socket leads to a delayed healing response13.

On account of these observations, a novel surgical technique was presented in literature (Caiazzo et al. 2010)14, with the name of Buccal Plate Augmentation (BPA). After performing a gentle tooth extraction and verifying the integrity of the alveolar walls, BPA consists in placing a HA-based bone graft material over the intact buccal bone plate, underneath the soft tissues and the periosteum in a surgically created pouch with the aim to maintain or augment crestal volumetry and soft tissue aesthetics of the region. This approach allows for avoiding recession of the alveolar facial wall without interfering with the natural healing mechanism of the extraction socket, which is left undisturbed. To date, however, there is still no evidence regarding the most suitable biomaterial for maintaining predictably crestal volumetry and soft tissues contour overtime.

ELIGIBILITY:
Inclusion Criteria:

* The local inclusion criteria are the following:

  1. indication for a tooth extraction in the incisor, canine or premolar area of the upper arch (for any clinical reason);
  2. presence of at least one tooth adjacent to the one to be extracted;
  3. presence of at least 5 mm. of vertical bone support around the tooth to be extracted;
  4. presence of an intact buccal plate in the extraction socket;
  5. age of the patient >18 years;
  6. patient will not wear any kind of removable prosthesis over the treatment area;
  7. patient will not undergo implant surgery in the treatment area up to 6 month from the extraction;
  8. patient willing and fully capable to comply with the study protocol;
  9. written informed consent given

Exclusion Criteria:

* acute myocardial infarction within the past 2 months,
* uncontrolled coagulation disorders,
* uncontrolled metabolic diseases (diabetes mellitus and bone pathologies),
* radiotherapy to the head/neck district within the past 24 months,
* present or past treatment with intravenous bisphosphonates,
* psychological or psychiatric problems, and alcohol or drugs abuse.
* Local exclusion criterion is the presence of uncontrolled or untreated periodontal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, DDS, Study Director — University of Trieste; Chiara O Navarra, DDS,PHD, Principal Investigator — University of Trieste; Roberto Di Lenarda, DDS, PHD, Study Chair — University of Trieste
Locations (1):
- University of Trieste, Trieste, TS, Italy